CLINICAL TRIAL: NCT01078675
Title: An Efficacy and 2-Year Safety Study of Open-label Rosuvastatin in Children and Adolescents (Aged From 6 to Less Than 18 Years) With Familial Hypercholesterolaemia
Brief Title: An Study to Evaluate Rosuvastatin in Children and Adolescents With Familial Hypercholesterolaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3561C00002
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Familial Hypercholesterolaemia
Keywords: Familial Hypercholesterolaemia; pediatric
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rosuvastatin calcium

INTERVENTIONS:
Drug: rosuvastatin calcium — 5 mg, oral, once daily, 24 months
  Other Names: Crestor
Drug: rosuvastatin calcium — 10 mg, oral, once daily, 24 months
  Other Names: Crestor
Drug: rosuvastatin calcium — 20 mg, oral, once daily, 24 months
  Other Names: Crestor

SUMMARY:
This study is being carried out to see if the study medication, rosuvastatin, is effective in treating familial hypercholesterolaemia in children and adolescents, and to determine the long term (over 2 years) safety, tolerability and efficacy of the study medication in these patients.

This study will also measure levels of drug in the blood and see how well it is tolerated. This is known as pharmacokinetic (PK) analysis.

At baseline only a small number of patients will participate in a single dose PK phase over 24 hours.

In order to see if this medication works, a control group of healthy siblings will help the researchers to compare certain results.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents (aged 6 to less than 18 years) with Familial Hypercholesterolaemia
* Patients aged between 6 and less than 10 years of age must not be taking a statin medicine

Exclusion Criteria:

* History of muscle or sensitivity reactions to any statin medicines
* Current active liver disease or dysfunction (except a confirmed diagnosis of Gilbert's disease)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J.P. Kastelein, MD, PhD, Principal Investigator — Chairman, Dept. of Vascular Medicine, Academic Medical Center, Meibergdreef 9
Locations (15):
- Research Site, Cincinnati, Ohio, United States
- Belgium (2):
  - Research Site, Leuven, Belgium
  - Research Site, Leuven
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec, Quebec
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Hoorn
  - Research Site, Leiderdorp
  - Research Site, Rotterdam
  - Research Site, Waalwijk
- Research Site, Oslo, Norway

REFERENCES:
- [Derived] Braamskamp MJAM, Langslet G, McCrindle BW, Cassiman D, Francis GA, Gagne C, Gaudet D, Morrison KM, Wiegman A, Turner T, Miller E, Kusters DM, Raichlen JS, Martin PD, Stein EA, Kastelein JJP, Hutten BA. Effect of Rosuvastatin on Carotid Intima-Media Thickness in Children With Heterozygous Familial Hypercholesterolemia: The CHARON Study (Hypercholesterolemia in Children and Adolescents Taking Rosuvastatin Open Label). Circulation. 2017 Jul 25;136(4):359-366. doi: 10.1161/CIRCULATIONAHA.116.025158. Epub 2017 Jun 7. PMID 28592434
- [Derived] Kusters DM, Wiegman A, Kastelein JJ, Hutten BA. Carotid intima-media thickness in children with familial hypercholesterolemia. Circ Res. 2014 Jan 17;114(2):307-10. doi: 10.1161/CIRCRESAHA.114.301430. Epub 2013 Nov 5. PMID 24192652
- [Derived] Tolani S, Pagler TA, Murphy AJ, Bochem AE, Abramowicz S, Welch C, Nagareddy PR, Holleran S, Hovingh GK, Kuivenhoven JA, Tall AR. Hypercholesterolemia and reduced HDL-C promote hematopoietic stem cell proliferation and monocytosis: studies in mice and FH children. Atherosclerosis. 2013 Jul;229(1):79-85. doi: 10.1016/j.atherosclerosis.2013.03.031. Epub 2013 Apr 19. PMID 23684512
- See also: D3561C00002 Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1357&filename=D3561C00002.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 250 patients with FH were screened. Additionally, 65 healthy siblings (HS) were enrolled. HS refers to healthy subjects that were siblings of either the study participants or other paediatric patients with HeFH that were not participating in the study. HS were enrolled to have assessments of cIMT, but did not participate further.
Groups:
- Rosuvastatin: Rosuvastatin 5 mg, 10 mg or 20 mg
- Healthy Siblings: Controls to HeFH patients in the cIMT evaluations
Period: Overall Study
Arm/Group | Rosuvastatin | Healthy Siblings
Started | 250 | 65
Patients Treated | 198 | 0
Completed | 182 | 59 (Healthy siblings did not participate in investigational product administration.)
Not Completed | 68 | 6
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Protocol Violation | 56 | 0
Not completed — Provided in CRF for specific reasons | 2 | 3
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Rosuvastatin; All treated patients. Healthy siblings; All patient who started this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Healthy Siblings | Total
Number analyzed (Participants) | 198 | 65 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 11.6 (3.33) | 11.5 (3.53) | 11.55 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 32 | 142
  Male | 88 | 33 | 121
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 178 | 53 | 231
  non-Caucasian | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C
Description: Negative values represent a decrease and positive values represent an increase. In total, 198 patients were treated. One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Time Frame: At Month 3, Month 12 and Month 24
Population: Intent-to-treat analysis set and Per-protocol analysis set
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Percentage change
  LDL-C %Change from Baseline at month 3 | -37.86 (14.392)
  LDL-C %Change from Baseline at month 12 | -43.67 (14.896)
  LDL-C %Change from Baseline at month 24 | -42.88 (18.222)
Statistical Analysis 1: Comparison: Rosuvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value<0.001 at Month 24. No adjustment for multiple comparisons is made for individual age group; P-value is two-sided and based on ANCOVA using age group as the fixed factor, and study centre and the baseline value as covariates; Mean Difference (Final Values) = -42.88, -42.88% CI 2-sided [-45.44 to -40.32], Standard Deviation 18.222

2. Primary Outcome: Sexual Maturation by Tanner Staging at Baseline
Description: Tanner stages (I-V) was used to characterize physical development in children and adolescent. The stages was based on external primary and secondary sex characteristics, such as the size of the breasts, genitalia, and development of pubic hair. Tanner stage is considered going up when the organs grow bigger.
Time Frame: At Baseline
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Participants
  Tanner Stage I at Baseline | 81 (NA)
  Tanner Stage II at Baseline | 32 (NA)
  Tanner Stage III at Baseline | 18 (NA)
  Tanner Stage IV at Baseline | 44 (NA)
  Tanner Stage V at Baseline | 21 (NA)
  Not Recorded at Baseline | 1

3. Primary Outcome: Single Dose PK - Cmax
Description: Serial plasma samples were taken at baseline (Week 0) at: 0.5 hours pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 9, 12 hours and on Day 1 at 24 hours after the single 10 mg dosing
Time Frame: Serial blood samples over 24 hours.
Population: Single dose PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Rosuvastatin: Rosuvastatin 10 mg
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 12
ng/mL | 3.5717 (3.22350)

4. Secondary Outcome: Percent Change From Baseline in HDL-C, TC, TG, Non-HDL-C, LDL-C/HDL-C, TC/HDL-C, Non HDL C/HDL-C, ApoB, ApoA-1, and ApoB/ApoA-1
Description: One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Time Frame: At Month 3, Month 12 and Month 24
Population: Intent-to-treat analysis set (LOCF)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Percent change
  HDL-C %Change from Baseline at Month 3 | 5.67 (17.445)
  HDL-C %Change from Baseline at Month 12 | 6.35 (16.725)
  HDL-C %Change from Baseline at Month 24 | 11.73 (19.996)
  TC %Change from Baseline at Month 3 | -29.60 (11.433)
  TC %Change from Baseline at Month 12 | -33.91 (12.050)
  TC %Change from Baseline at Month 24 | -32.03 (14.530)
  Triglycerides %Change from Baseline at Month 3 | -7.95 (34.482)
  Triglycerides %Change from Baseline at Month 12 | -7.85 (37.530)
  Triglycerides %Change from Baseline at Month 24 | -0.12 (37.682)
  non-HDL C %Change from Baseline at Month 3 | -36.35 (13.368)
  non-HDL C %Change from Baseline at Month 12 | -41.66 (14.235)
  non-HDL C %Change from Baseline at Month 24 | -40.40 (17.555)
  LDL-C/HDL-C %Change from Baseline at Month 3 | -39.66 (17.381)
  LDL-C/HDL-C %Change from Baseline at Month 12 | -45.63 (17.082)
  LDL-C/HDL-C %Change from Baseline at Month 24 | -46.95 (20.126)
  TC/HDL-C %Change from Baseline at Month 3 | -31.77 (14.874)
  TC/HDL-C %Change from Baseline at Month 12 | -36.54 (14.474)
  TC/HDL-C %Change from Baseline at Month 24 | -37.39 (17.079)
  Trig/HDL-C %Change from Baseline at Month 3 | -9.05 (41.765)
  Trig/HDL-C %Change from Baseline at Month 12 | -10.50 (40.633)
  Trig/HDL-C %Change from Baseline at Month 24 | -7.12 (40.585)
  non-HDL-C/HDL-C %Change from Baseline at Month 3 | -37.98 (17.369)
  non-HDL-C/HDL-C %Change from Baseline at Month 12 | -43.71 (16.731)
  non-HDL-C/HDL-C %Change from Baseline at Month 24 | -44.74 (19.896)
  ApoA-I %Change from Baseline at Month 3 | 4.77 (14.680)
  ApoA-I %Change from Baseline at Month 12 | 1.41 (13.747)
  ApoA-I %Change from Baseline at Month 24 | 2.34 (15.027)
  ApoB %Change from Baseline at Month 3 | -29.29 (12.456)
  ApoB %Change from Baseline at Month 12 | -35.65 (12.424)
  ApoB %Change from Baseline at Month 24 | -35.72 (15.710)
  ApoB/ApoA-I %Change from Baseline at Month 3 | -31.30 (15.524)
  ApoB/ApoA-I %Change from Baseline at Month 12 | -35.66 (13.920)
  ApoB/ApoA-I %Change from Baseline at Month 24 | -35.94 (18.743)
  hsCRP %Change from Baseline at Month 3 | 512.57 (4724.249)
  hsCRP %Change from Baseline at Month 12 | 42.96 (226.954)
  hsCRP %Change from Baseline at Month 24 | 98.36 (565.444)

5. Secondary Outcome: Change From Baseline in Max and Mean Carotid Intima and Media Wall Thickness (cIMT)
Description: as for outcome 4
Time Frame: At Month 12 and Month 24
Population: Intent-to-treat analysis set (LOCF) and healthy siblings
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rosuvastatin | Healthy Siblings
Number analyzed (Participants) | 197 | 65
mm
  Max cIMT Change from Baseline at Month 12 | 0.00626 (0.073446) | 0.01707 (0.056223)
  Max cIMT Change from Baseline at Month 24 | 0.00189 (0.060864) | 0.01202 (0.049102)
  Mean cIMT Change from Baseline at Month 12 | 0.00282 (0.041186) | 0.01564 (0.032052)
  Mean cIMT Change from Baseline at Month 24 | 0.01056 (0.040762) | 0.02779 (0.031004)

6. Secondary Outcome: Adverse Events
Description: Number of participants with Various Categories of AE's. One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Time Frame: 2-year study period
Population: Safety analysis set
Measure: Number; unit: Participant
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Participant
  Any AE | 172
  AE Leading to Death | 0
  AE Leading to Discontinuation | 3
  Serious AE | 9
  Treatment Related AE | 29
  Treatment Related AE Leading to Death | 0
  Treatment Related AE Leading to Discontinuation | 3
  Treatment Related Serious AE | 0

7. Secondary Outcome: Total Duration of Exposure
Description: Total duration of exposure was calculated as [last dose date of rosuva - first dose date of rosuva + 1 day]. One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Time Frame: 2-year study period
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Days | 703.5 (97.25)

8. Primary Outcome: Percent Change From Baseline in Height
Description: as for outcome 4
Time Frame: At Month 12 and Month 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Percent change
  %Change from Baseline at Month 12 | 3.20 (2.023)
  %Change from Baseline at Month 24 | 5.91 (3.968)

9. Primary Outcome: Sexual Maturation by Tanner Staging at Month 12
Description: as for outcome 2
Time Frame: At Baseline
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Participants
  Tanner Stage I at Month 12 | 61 (NA)
  Tanner Stage II at Month 12 | 31 (NA)
  Tanner Stage III at Month 12 | 21 (NA)
  Tanner Stage IV at Month 12 | 32 (NA)
  Tanner Stage V at Month 12 | 42 (NA)
  Not Recorded at Month 12 | 10

10. Primary Outcome: Sexual Maturation by Tanner Staging at Month 24
Description: as for outcome 2
Time Frame: At Baseline
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Participants
  Tanner Stage I at Month 24 | 43 (NA)
  Tanner Stage II at Month 24 | 33 (NA)
  Tanner Stage III at Month 24 | 23 (NA)
  Tanner Stage IV at Month 24 | 32 (NA)
  Tanner Stage V at Month 24 | 64 (NA)
  Not Recorded at Month 24 | 2

11. Primary Outcome: Single Dose PK - Tmax
Description: as for outcome 3
Time Frame: Serial blood samples over 24 hours
Population: Single dose PK analysis set
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 12
hr | 2.664 (1.8851)

12. Primary Outcome: Single Dose PK - AUC(0-24)
Description: as for outcome 3
Time Frame: Serial blood samples over 24 hours
Population: Single dose PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 12
ng*hr/mL | 27.675 (26.6417)

13. Secondary Outcome: Overal Treatment Adherence
Description: Overall adherence rate was calculated as the weighted mean of adherence rates of all consecutive visits after baseline, in which the adherence rate between 2 consecutive visits was a percentage of the number of rosuvastatin taken divided by duration of exposure. One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Time Frame: 2-year study period
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Percent of doses
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 197
Percent of doses | 89.6 (12.25)

ADVERSE EVENTS:
Time Frame: Treatment Phase
Description: One patient received 1 dose of study drug but was not included in the efficacy and safety analyses due to a lack of follow-up data.
Arm/Group | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 9/197
Other Adverse Events (participants affected / at risk) | 172/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=197)
Appendicitis (Infections and infestations) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Streptococcal toxic shock syndrome (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Leg fracture (Injury, poisoning and procedural complications) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (2)
Pectus carinatum (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=197)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Pectus carinatum (Congenital, familial and genetic disorders) | 1 (2)
Auricular swelling (Ear and labyrinth disorders) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 2 (2)
Early menarche (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (18)
Abdominal pain upper (Gastrointestinal disorders) | 15 (21)
Constipation (Gastrointestinal disorders) | 4 (4)
Dental discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 4 (6)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (24)
Rectal spasm (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 19 (24)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (8)
Influenza like illness (General disorders) | 16 (19)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 10 (10)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 4 (4)
Seasonal allergy (Immune system disorders) | 4 (4)
Amoebic dysentery (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 3 (5)
Ear infection (Infections and infestations) | 4 (5)
Eye infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 12 (15)
Gastroenteritis viral (Infections and infestations) | 18 (24)
Gingival infection (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 3 (3)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 20 (28)
Laryngitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Mononucleosis syndrome (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 88 (150)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 3 (3)
Pertussis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 8 (10)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (4)
Tonsillitis (Infections and infestations) | 4 (6)
Tooth infection (Infections and infestations) | 2 (2)
Toxic shock syndrome streptococcal (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (12)
Urinary tract infection (Infections and infestations) | 7 (7)
Viral infection (Infections and infestations) | 2 (2)
Viral pericarditis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (2)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (5)
Cardiac murmur (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (2)
Lymphocyte count abnormal (Investigations) | 1 (1)
Renal bruit (Investigations) | 1 (1)
Serum ferritin decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 2 (4)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 6 (8)
Epilepsy (Nervous system disorders) | 1 (4)
Headache (Nervous system disorders) | 46 (76)
Migraine (Nervous system disorders) | 3 (11)
Paraesthesia (Nervous system disorders) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 6 (11)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2)
Autism spectrum disorder (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (2)
Pyuria (Renal and urinary disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Xanthoma (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No